CLINICAL TRIAL: NCT01227499
Title: Differential Diagnosis Value of Peak Systolic Velocity of Thyroid Superior Artery Using Color Flow Doppler Sonography in Transient Thyrotoxicosis Caused by Thyroiditis and Graves Disease
Brief Title: Differential Diagnosis of STA-PSV in Thyrotoxicosis
Status: Completed | Type: Observational
Sponsor: xiaolong zhao (Other)
Collaborators: Zhongda Hospital (Other); Fudan University (Other)
Responsible Party: Sponsor-Investigator, xiaolong zhao, endocrinology department, Huashan Hospital
Organization: Huashan Hospital (Other)
Other Study IDs: huashan001
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Thyrotoxicosis; Peak Systolic Velocity of Superior Thyroid Artery; Thyroiditis; Graves Disease
MeSH Terms: conditions — Thyrotoxicosis; Thyroiditis; Graves Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Aim: Graves's disease and thyroiditis can both characterized with thyrotoxicosis, but their clinical outcome and therapy is quiet different. Measurement of iodine uptake is the gold standard to differential diagnosis the thyroiditis or Graves's disease. But the iodine uptake is limited for its availability in china and easily influenced by medicine or food contained iodine.The blood pattern of thyroid CFDS is useful for differentiate the cause of thyrotoxicosis.Most previous studies using the descriptive pattern of thyroid CFDS is easily varied by operator subjective judgement. This study is focus on the role of peak systolic velocity of thyroid superior artery in differential diagnosis of thyrotoxicosis. Methods: Patients with thyrotoxicosis symptoms without recent medicine history were enrolled in two clinical center. Its thyroid function, iodine uptake , CFDS of thyroid and peak systolic velocity of thyroid superior artery is detected. Thyrotoxicosis is defined as TSH level below the low value of normal range. Graves disease is defined as the typical symptoms of graves disease such as graves ophthalmopathy or increased iodine uptake. Thyroiditis is defined as lack of typical symptoms of graves disease or decreased iodine uptake.We use receiver operator curve(ROC) to evaluate its diagnosis value

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed without taking any antithyroid drug or beta receptor blocker with TSH level below the lower limits of reference range
* is willing to be enrolled

Exclusion Criteria:

* unwilling
* taking antithyroid drug or beta receptor blocker
* taking foods or medicine rich in iodine in 8 weeks
* women with pregnant or lactation

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
mean STA-PSV | 2014-04-07
  the mean STA-PSV
uptake of iodine | December 1, 2013

SECONDARY OUTCOMES:
PSV | December 1, 2013

OTHER OUTCOMES:
thyroid funciton | December 1, 2013

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaolong Zhao, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Zhao X, Chen L, Li L, Wang Y, Wang Y, Zhou L, Zeng F, Li Y, Hu R, Liu H. Peak systolic velocity of superior thyroid artery for the differential diagnosis of thyrotoxicosis. PLoS One. 2012;7(11):e50051. doi: 10.1371/journal.pone.0050051. Epub 2012 Nov 16. PMID 23166817